CLINICAL TRIAL: NCT07102966
Title: MAGNET: Making Genomics Accessible For Newborns In Texas
Brief Title: Genetic Study to Determine the Cause of Birth Defects in Newborns in Texas
Acronym: MAGNET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Seema Lalani, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-56296; 1R01HG013428-01A1 (NIH)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Rare Diseases
Keywords: Rapid whole genome sequencing, newborns, Texas
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAGNET study patients (Experimental): Patients receiving rapid whole genome sequencing
  Interventions: Genetic: Rapid whole genome sequencing

INTERVENTIONS:
Genetic: Rapid whole genome sequencing — All consented patients will receive a virtual genetic evaluation and rapid whole genome sequencing

SUMMARY:
The purpose of this study is to provide advanced genetic testing and virtual consultations for seriously ill newborns in hospitals in Texas with fewer resources, especially along the Texas-Mexico border. The researchers also want to know how well the virtual consultation tool, called Consultagene, works in these hospitals by gathering feedback from healthcare providers. Researchers will provide rapid whole genome sequencing (WGS) to 200 infants over a period of 5 years. Data will be collected via Consultagene, surveys, and qualitative interviews.

DETAILED DESCRIPTION:
The study will use advanced testing such as WGS and RNA sequencing to look for possible diagnoses in infants. Only newborns with an unknown genetic diagnosis and admitted to a NICU in select Texas hospitals will be included. The researchers have executed broad reliance agreements with the participating NICUs in the study. Baylor IRB will serve as the IRB of record for all participating sites. All referrals will be received through Consultagene (www.consultagene.org).

Baylor College of Medicine (BCM) will conduct virtual genetic evaluations using video visits, with help from the local hospital team. Photos and medical records will be reviewed, and blood or buccal swabs will be collected from the infants and parents. Test results will be returned in about a week, and researchers will provide genetic counseling to families through another virtual visit. If needed, additional testing will be done. Families will be connected to support groups, treatment options, and clinical trials if available.

To understand the impact of the study, families will be asked to complete two short surveys; one at the beginning and one after they receive results. Doctors who use Consultagene will also be surveyed and interviewed to learn about their experience and gather feedback for improving the virtual tool.

All data will be kept private and secure. DNA samples collected will be stored at BCM for future research, but without any identifying information. Samples may also be shared with other researchers studying similar health conditions, but only under strict guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Undiagnosed infants from 0-90 days of age, with a diverse group of phenotypes and strongly suspected to have genetic disorders.

Exclusion Criteria:

* (1) abnormal noninvasive prenatal testing (NIPT) suggesting chromosomal abnormality; (2) abnormal amniocentesis results, (3) abnormal newborn screening indicating an inborn error of metabolism; (4) abnormal FISH results for aneuploidy (trisomy 18, 13, or monosomy X); (5) Down syndrome; (6) dysmorphic features in the absence of other congenital anomalies; (7) isolated birth defects such as myelomeningocele, cleft lip/palate, cardiac septal defects, isolated congenital diaphragmatic hernia, etc.; (8) birth defects due to known teratogens i.e., alcohol, Isotretinoin, etc.; (9) multiple congenital anomalies associated with maternal diabetes; (10) VACTERL association; and (11) hemodynamically unstable newborns needing transport for higher level of care.

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 410 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Consultagene | From enrollment to the end of treatment-4 years
  The primary outcome will be effectiveness of Consultagene, defined as difference in diagnostic yield compared to usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Lee, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Unending (Beginning 1 year after publication with no end date)

REFERENCES:
- [Background] Vuocolo B, Sierra R, Brooks D, Holder C, Urbanski L, Rodriguez K, Gamez JD, Mulukutla SN, Hernandez A, Allegre A, Hidalgo H, Rodriguez S, Magallan S, Gibson J, Bernini JC, Watson M, Nelson R, Mellin-Sanchez L, Garcia N, Berry L, Dai H, Soler-Alfonso C, Carter K, Lee B, Lalani SR. Project GIVE: using a virtual genetics service platform to reduce health inequities and improve access to genomic care in an underserved region of Texas. J Neurodev Disord. 2024 Sep 9;16(1):52. doi: 10.1186/s11689-024-09560-x. PMID 39251895

DOCUMENTS (1):
  • Study Protocol (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT07102966/Prot_000.pdf